CLINICAL TRIAL: NCT02121600
Title: Assessment of CRPC Response Through Comprehensive Characterization Using Novel Biomarkers (PET CRPC)
Brief Title: 18F-FCH PET/MRI to Assess Tumor Response in Castration Resistant Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PET CRPC
Record Dates: First submitted 2014-04-15; First posted 2014-04-23 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Prostate Cancer
Keywords: Fluorocholine (FCH); Positron Emission Tomography (PET); Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel (Other): Patients who will be receiving Docetaxel as cancer treatment will be assigned to Arm 1. All patients in this cohort will have a [F-18]-FCH PET scan with full body MRI scan
  Interventions: Other: [F-18]-FCH; Radiation: PET scan; Radiation: MRI scan
- Abiraterone (Other): Patients who will be receiving Abiraterone as cancer treatment will be assigned to Arm 2. All patients in this cohort will have a [F-18]-FCH PET scan with full body MRI scan.
  Interventions: Other: [F-18]-FCH; Radiation: PET scan; Radiation: MRI scan

INTERVENTIONS:
Other: [F-18]-FCH — Before the PET/MRI or PET/CT scan, patients will receive an [F-18]-Fluorocholine injection in the arm.
  Other Names: [F-18]-Fluorocholine Injection
Radiation: PET scan — A whole body PET scan will be performed, combined with either whole body MRI or CT scan. This will be performed at baseline and after 12 weeks of treatment
Radiation: MRI scan — Whole body MRI scan will be performed. This may be combined with PET scan or may be performed separately. MRI scan will be done at baseline and after 12 weeks of treatment

SUMMARY:
Evaluate the ability of 18F-FCH PET/MRI scan to detect pre-treatment tumor burden and assess response to treatment in men with castration resistant prostate cancer (CRPC).

It is hypothesized that these novel biomarkers will better identify evaluable lesions prior to therapy and identify response to treatment (or lack thereof) earlier in the treatment period, providing a better guide for treating men with CRPC.

DETAILED DESCRIPTION:
Castrate resistant prostate cancer (CRPC) occurs when prostate cancer no longer responds to androgen deprivation therapy. Eventually all men diagnosed with CRPC will succumb to their disease. While many new therapies have been introduced, there are limitations in assessing treatment response and physicians are faced with a challenge when creating a management strategy for men with CRPC.

Most men present with bone metastases, and accurate quantification of disease burden can be difficult due to the nature of conventional scans such as CT and bone scan. In addition, the standard blood PSA measurement does not always reflect a clinical response, or may lag to show this response. There is a clear need for better imaging and blood biomarkers to measure disease in men with CRPC.

This study will explore the benefit of a 18F-FCH Hybrid PET/MRI scan, Cancer Microparticle (CMP) and Circulating Tumor Cell (CTC) measurements compared to standard imaging and PSA levels.

In this study, patients will receive a 18F-FCH PET/MRI or 18F-FCH PET/CT scan + whole body MRI at baseline and after 12 weeks of treatment. Serial CMP and CTC blood samples will be taken at 5 study timepoints.

66 patients will be enrolled at 3 cancer centres in Ontario. Patients will be divided into 2 cohorts based on the type of treatment they will receive: Docetaxel or Abiraterone.

It is hypothesized that these novel biomarkers will better identify evaluable lesions prior to therapy and identify response to treatment (or lack thereof) earlier in the treatment period thus providing a better guide for treating men with CRPC.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patient with CRPC and experiencing disease progression as defined by PCWG2
* ECOG 0-2
* Must continue gonadal castrative therapy
* Has completed antiandrogen withdrawal ≥ 6 weeks prior to registration
* Metastatic disease documented by imaging
* Patient is planned for treatment with docetaxel or abiraterone
* If treated with bisphosphonates or denosumab, has been on these for ≥ 6 weeks.
* Must provide written informed consent

Exclusion Criteria:

* Prior history of invasive malignant disease unless disease free for at least 5 years, with the exception of non-melanoma skin cancer
* Planned for any concurrent anticancer treatment oher than docetaxel or abiraterone
* Prior radiotherapy or surgery within 4 weeks of start of docetaxel or abiraterone
* Inability to comply with the imaging requirements (eg. inability to lie supine for one hour)
* Allergy to MRI contrast agent or PET tracer to be used as part of the imaging
* Sickle cell disease or other hemoglobinopathies
* Insufficient renal function (eGFR ≤ 30 mL/min)
* Known residual bladder volume > 150 cc
* Hip prosthesis or intrabdominal vascular grafting
* Contraindication to CT contrast
* Contraindication to MRI as per institutional policy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-09; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Number of lesions detected with 18F-FCH PET/MRI compared to conventional imaging | 3 years

SECONDARY OUTCOMES:
Number of concordant lesions identified on identified on 18F-FCH PET, conventional imaging and MRI | 3 years
Concordance between number Circulating Tumor Cells (CTCs) and Cancer Microparticles (CMPs) and number of lesions detected by PET/MRI and conventional imaging | 3 years
  At both baseline and after 12 weeks of treatment
Change in number and size of lesions after 12 weeks of treatment | 3 years
  As detected by 18F-FCH PET/MRI and change in CTC and CMP values
Progression Free Survival | 6 years
  Changes in lesion parameters on PET and MRI and changes in serial CTC and CMP levels will be assessed to see if they are predictive of progression free survival
Overall Survival | 6 years
  Changes in lesion parameters on PET and MRI and changes in serial CTC and CMP levels will be assessed to see if they are predictive of overall survival

OTHER OUTCOMES:
Percentage of change in clinical management based on results of 18F-FCH PET/MRI and CTC results | 3 years
Concordance of identified lesions on hybrid PET/CT + fused MRI vs hybrid PET/MRI | 3 years
Concordance between CTC values on a new microfluidics-based CTC assay and the FDA/Health Canada approved CellSearch CTC assay (clinical gold standard) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Winquist, MD, Principal Investigator — London Health Sciences Centre
Locations (3):
- Canada (3):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario